CLINICAL TRIAL: NCT01784627
Title: Randomized Controlled Trial of Computerized SBI to Reduce Teen Alcohol Use
Brief Title: Trial of Computerized SBI to Reduce Teen Alcohol Use
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No funding
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, John R Knight, MD, Associate Professor of Pediatrics, Harvard Medical School; Senior Associate in Medicine; Associate in Psychiatry, Director, Center for Adolescent Substance Abuse Research, Boston Children's Hospital, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JK R01 PA-12-031
Record Dates: First submitted 2013-02-04; First posted 2013-02-06 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Alcohol Abuse; Cannabis Abuse; Nicotine Dependence
Keywords: substance use; alcohol abuse; cannabis abuse; nicotine dependence; adolescents
MeSH Terms: conditions — Alcoholism; Marijuana Abuse; Tobacco Use Disorder; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment at Usual (No Intervention): Participants in this group will receive treatment as usual (TAU) from their provider, which may or may not include screening and brief advice regarding alcohol use.
- c-ASBI (Experimental): Participants in this group will receive the computerized alcohol screening and brief intervention (c-ASBI).
  Interventions: Behavioral: c-ASBI

INTERVENTIONS:
Behavioral: c-ASBI — Participants in the c-ASBI group will complete a computerized screen for alcohol, cannabis, tobacco and other drugs, then view their screen score and 10 pages of information about the health effects of substance use and true-life stories on the computer. Their provider will see a report of their screen results and provide advice to stop or decrease their use, or, for those at high risk, referral to complete a computerized motivational enhancement therapy intervention.
  Arms: c-ASBI

SUMMARY:
The goal of this project is to test the effectiveness of a computer-facilitated alcohol screening and brief intervention (c-ASBI) system for 12- to 18-year-old primary care patients in a multi-site, randomized comparative effectiveness trial. The investigators hypothesize that, among 12- to 18-year olds patients coming for annual well-care, those receiving c-ASBI will have lower rates of any alcohol use at 3-, 6-, and 12-month follow-ups compared to Treatment As Usual (TAU).

DETAILED DESCRIPTION:
The Specific Aims are to 1) Test the effects of c-ASBI on any alcohol use; 2) Test the effects of c-ASBI separately as a prevention, therapeutic, and risk-reduction intervention; 3) Test the effects of c-ASBI separately on cannabis and tobacco use; explore its effects on other drug use; and 4) Assess potential moderators (e.g., age, gender, race/ethnicity, substance use history +/-, parent/sibling/peer substance use), mediators (e.g., Youth to Provider Connectedness,20 perceived harmfulness of alcohol and drug use), and explore c-ASBI's mechanism of action.

ELIGIBILITY:
Inclusion Criteria:

* Arriving for well or non-emergent care at one of participating study sites
* Have an email address
* Have internet address

Exclusion Criteria:

* Unable to read or understand English
* Living away at college at the time of the recruitment visit
* Not available for computer/telephone follow-ups
* Judged by the provider to be medically or emotionally unstable at time of visit

Ages: 9 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Days of alcohol use | 12 months
  We will compare rates of any alcohol use over the past twelve months between the groups.

SECONDARY OUTCOMES:
Drinking initiation | 12 months
  We will compare rates of drinking initiation over the past 12-months between groups.
Drinking cessation | 12 months
  We will compare rates of drinking cessation over the past 12 months between groups.
Driving/Riding risk | 12 months
  We will compare the rates of driving under the influence or riding with a driver under the influence between groups.

OTHER OUTCOMES:
Cannabis use | 12 months
  We will compare the rates of cannabis use over the past twelve months between groups.
Tobacco use | 12 months
  We will compare the rates of tobacco use over the past twelve months between groups.

CONTACTS AND LOCATIONS:
Overall Officials: John R Knight, MD, Principal Investigator — Boston Children's Hospital
Locations (6):
- United States (6):
  - Tufts Medical Center, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Longwood Pediatrics, Boston, Massachusetts
  - East Boston Neighborhood Health Center, Boston, Massachusetts
  - Cambridge Pediatrics, Cambridge, Massachusetts
  - Lexington Pediatrics, Lexington, Massachusetts

IPD SHARING:
Plan to Share IPD: No